CLINICAL TRIAL: NCT00887328
Title: Extending the Time for Thrombolysis in Emergency Neurological Deficits
Acronym: EXTEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government); University of Melbourne (Other); Melbourne Health (Other); The Florey Institute of Neuroscience and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTA0901
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: ischemic stroke; ischemic penumbra; magnetic resonance imaging; MRI; diffusion imaging; DWI; perfusion imaging; PWI; thrombolysis; alteplase; tPA; EPITHET
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV tPA (Experimental): intravenous tissue plasminogen activator
  Interventions: Drug: Tissue Plasminogen Activator (Alteplase)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tissue Plasminogen Activator (Alteplase) — 0.9 mg/kg up to a maximum of 90mg, intravenous, 10% as bolus and the remainder over 1 hour
  Other Names: Actilyse; Activase; tPA; r-tPA
  Arms: IV tPA
Drug: Placebo — placebo provided as 50mg lyophilised powder to be reconstituted with sterile water in glass vials indistinguishable from active drug
  Arms: Placebo

SUMMARY:
The primary hypothesis being tested in this trial is that ischaemic stroke patients selected with significant penumbral mismatch (measured by MRI criteria) at 3 - 9 hours post onset of stroke will have improved clinical outcomes when given intravenous tissue plasminogen activator (tPA) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with hemispheric acute ischaemic stroke
2. Patient, family member or legally responsible person depending on local ethics requirements has given informed consent
3. Patient's age is ≥18 years
4. Treatment onset can commence within ≥ 3 - 9 hours after stroke onset according to registered product information, or within 4.5 - 9 hours according to locally accepted guidelines*.

   (*Guidelines are currently under international review - advisory statement issued by the Stroke Council, American Heart Association and American Stroke Association)
5. Patients who wake with stroke may be included if neurological and other exclusion criteria are satisfied. These 'wake up' strokes are defined as having no symptoms at sleep onset, but stroke symptoms on waking. The time of stroke onset is to be taken as the mid-point between sleep onset (or last known to be normal) and time of waking. The maximum time window for randomisation is then 9 hours from the mid-point as described.
6. NIHSS score of ≥ 4 - 26 with clinical signs of hemispheric infarction.
7. Penumbral mismatch - A "hypo-perfusion to core" volume ratio of greater than 1.2 and an absolute difference greater than 10mL (using a MR or CT Tmax > 6 second delay) between perfusion lesion and MR-DWI or CT-CBF core lesion.
8. An ischaemic core lesion volume of less than or equal to 70 ml using MR-DWI or CT-CBF ** Patients may be consented before or after penumbral screening depending upon local practice. The entire cohort of patients consented onto the study will be followed up with clinical assessments and biomarker studies regardless of eligibility for randomisation to treatment based on penumbral mismatch criteria

Exclusion Criteria:

1. Intracranial haemorrhage (ICH) identified by CT or MRI
2. Rapidly improving symptoms, particularly if in the judgment of the managing clinician that the improvement is likely to result in the patient having an NIHSS score of < 4 at randomization
3. Pre-stroke MRS score of ≥ 2 (indicating previous disability)
4. Contra indication to imaging with MR with contrast agents
5. Infarct core >1/3 MCA territory qualitatively
6. Participation in any investigational study in the previous 30 days
7. Any terminal illness such that patient would not be expected to survive more than 1 year
8. Any condition that could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study (this applies to patients with severe microangiopathy such as haemolytic uremic syndrome or thrombotic thrombocytopenic purpura). The judgment is left to the discretion of the Investigator.
9. Pregnant women (clinically evident)
10. Previous stroke within last three months
11. Recent past history or clinical presentation of ICH, subarachnoid haemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm. At the discretion of each Investigator.
12. Current use of oral anticoagulants or a prolonged prothrombin time (INR > 1.7) if the patient is on warfarin
13. Use of heparin, except for low dose subcutaneous heparin, in the previous 48 hours and an activated prolonged partial thromboplastin time exceeding the upper limit of the local laboratory normal range.
14. Use of glycoprotein IIb - IIIa inhibitors within the past 72 hours. Use of single or dual agent oral platelet inhibitors (clopidogrel and/or low-dose aspirin) prior to study entry is permitted.
15. Clinically significant hypoglycaemia.
16. Uncontrolled hypertension defined by a blood pressure > 185 mmHg systolic or >110 mmHg diastolic on at least 2 separate occasions at least 10 minutes apart, or requiring aggressive treatment to reduce the blood pressure to within these limits. The definition of "aggressive treatment" is left to the discretion of the responsible Investigator.
17. Hereditary or acquired haemorrhagic diathesis
18. Gastrointestinal or urinary bleeding within the preceding 21 days
19. Major surgery within the preceding 14 days which poses risk in the opinion of the investigator.
20. Exposure to a thrombolytic agent within the previous 72 hours
21. Clinically deemed eligible for Endovascular Clot Retrieval (ECR) treatment by the treating team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-06; Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) 0-1 | 3 months

SECONDARY OUTCOMES:
Categorical shift in modified Rankin Score (mRS) | 3 months
Change in ≥ 8 NIHSS points or reaching ≤ 1 on this scale | 3 months
Death due to any cause | 3 months
Symptomatic ICH | 24 hours
  Symptomatic hemorrhage defined by SITS-MOST criteria: type 2 parenchymal hematoma associated with ≥4 point increase in NIHSS
Reperfusion | 24 hours
Recanalisation | 24 hours
Infarct growth | 24 hours
  Difference in volumetric DWI volume between baseline and 24 hour MRI
Recurrent stroke | 3 and 12 months
Depression (Montgomery-Asberg Depression Rating Scale [MADRS]) | 3 and 12 months
Quality of life (Stroke Impact Scale) | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Donnan, MD FRACP, Principal Investigator — The Florey Institute of Neuroscence and Mental Health; Stephen Davis, MD FRACP, Principal Investigator — University of Melbourne
Locations (22):
- Australia (20):
  - Gosford Hospital, Kanwal, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Sunshine Coast University Hospital, Nambour, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Western Hospital, Footscray, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Helsinki University Central Hospital, Helsinki, Finland
- Auckland Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Bivard A, Churilov L, Ma H, Levi C, Campbell B, Yassi N, Meretoja A, Zhao H, Sharma G, Chen C, Davis S, Donnan G, Yan B, Parsons M; EXTEND investigators. Does variability in automated perfusion software outputs for acute ischemic stroke matter? Reanalysis of EXTEND perfusion imaging. CNS Neurosci Ther. 2022 Jan;28(1):139-144. doi: 10.1111/cns.13756. Epub 2021 Nov 16. PMID 34786868
- [Derived] Goodin P, Lamp G, Vidyasagar R, Connelly A, Rose S, Campbell BCV, Tse T, Ma H, Howells D, Hankey GJ, Davis S, Donnan G, Carey LM. Correlated Resting-State Functional MRI Activity of Frontostriatal, Thalamic, Temporal, and Cerebellar Brain Regions Differentiates Stroke Survivors with High Compared to Low Depressive Symptom Scores. Neural Plast. 2019 Jul 28;2019:2357107. doi: 10.1155/2019/2357107. eCollection 2019. PMID 31467520
- [Derived] Ma H, Campbell BCV, Parsons MW, Churilov L, Levi CR, Hsu C, Kleinig TJ, Wijeratne T, Curtze S, Dewey HM, Miteff F, Tsai CH, Lee JT, Phan TG, Mahant N, Sun MC, Krause M, Sturm J, Grimley R, Chen CH, Hu CJ, Wong AA, Field D, Sun Y, Barber PA, Sabet A, Jannes J, Jeng JS, Clissold B, Markus R, Lin CH, Lien LM, Bladin CF, Christensen S, Yassi N, Sharma G, Bivard A, Desmond PM, Yan B, Mitchell PJ, Thijs V, Carey L, Meretoja A, Davis SM, Donnan GA; EXTEND Investigators. Thrombolysis Guided by Perfusion Imaging up to 9 Hours after Onset of Stroke. N Engl J Med. 2019 May 9;380(19):1795-1803. doi: 10.1056/NEJMoa1813046. PMID 31067369
- [Derived] Churilov L, Ma H, Campbell BC, Davis SM, Donnan GA. Statistical Analysis Plan for EXtending the time for Thrombolysis in Emergency Neurological Deficits (EXTEND) trial. Int J Stroke. 2020 Feb;15(2):231-238. doi: 10.1177/1747493018816101. Epub 2018 Dec 7. PMID 30523735
- [Derived] Tse T, Binte Yusoff SZ, Churilov L, Ma H, Davis S, Donnan GA, Carey LM; START research team. Increased work and social engagement is associated with increased stroke specific quality of life in stroke survivors at 3 months and 12 months post-stroke: a longitudinal study of an Australian stroke cohort. Top Stroke Rehabil. 2017 Sep;24(6):405-414. doi: 10.1080/10749357.2017.1318339. Epub 2017 Apr 24. PMID 28438076